CLINICAL TRIAL: NCT04263038
Title: Clinical Surveillance vs. Anticoagulation for Low-risk Patients With Isolated Subsegmental Pulmonary Embolism: a Multicenter Randomized Placebo-controlled Non-inferiority Trial
Brief Title: Clinical Surveillance vs. Anticoagulation for Low-risk Patients With Isolated Subsegmental Pulmonary Embolism
Acronym: SAFE-SSPE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Drahomir Aujesky (Other)
Collaborators: University of Bern (Other); Schweizerischer Nationalfonds (Other); Leiden University Medical Center (Other); The Ottawa Hospital (Other); Bayer (Industry)
Responsible Party: Sponsor-Investigator, Drahomir Aujesky, Prof. Dr., MD, MSc, Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-02297
Record Dates: First submitted 2020-02-04; First posted 2020-02-10 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Embolism; Embolism; Embolism and Thrombosis; Lung Diseases; Cardiovascular Diseases; Respiratory Tract Diseases; Venous Thromboembolism; Anticoagulant-induced Bleeding; Bleeding
Keywords: subsegmental pulmonary embolism
MeSH Terms: conditions — Pulmonary Embolism; Embolism; Embolism and Thrombosis; Lung Diseases; Cardiovascular Diseases; Respiratory Tract Diseases; Venous Thromboembolism; Hemorrhage | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anticoagulation (Active Comparator): Patients in the anticoagulation group will receive rivaroxaban 15 mg twice daily for the first 21 days, followed by 20 mg once daily for an overall treatment duration of 90 days.
  Interventions: Drug: Rivaroxaban
- No anticoagulation (Placebo Comparator): Patients in the group without anticoagulation will receive placebo twice daily for the first 21 days, followed by one tablet daily for an overall treatment duration of 90 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rivaroxaban — Anticoagulation
  Arms: Anticoagulation
Drug: Placebo — Study drug without active agent
  Arms: No anticoagulation

SUMMARY:
The clinical significance of pulmonary embolism (PE) limited to the subsegmental pulmonary arteries, so called isolated subsegmental pulmonary embolism (SSPE), remains controversial. Whether isolated SSPE represents "true" PE, a clinically more benign form of PE, a physiologic lung clearing process, or a false positive result (artifact) is currently unclear and hence, whether patients with isolated SSPE benefit from anticoagulant treatment is uncertain. Despite growing evidence from observational studies that withholding anticoagulation may be a safe option in selected patients with isolated SSPE (i.e., those without concomitant deep vein thrombosis, cancer, etc.), most patients with isolated SSPE receive anticoagulant treatment, which is associated with an increased risk of bleeding. The overall objective of the randomized controlled SAFE-SSPE trial is to evaluate the efficacy and safety of clinical surveillance without anticoagulation compared to anticoagulation treatment in low-risk patients with isolated SSPE.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent as documented by signature
2. Age ≥18 years
3. Objective diagnosis of symptomatic or asymptomatic isolated SSPE

Exclusion Criteria:

1. Presence of leg deep vein thrombosis (DVT) or upper extremity DVT (subclavian vein or above)
2. Active cancer, defined as cancer treated with surgery, chemotherapy, radiotherapy, or palliative care during the last 6 months
3. ≥1 prior episode of unprovoked VTE (absence of a transient or permanent risk factor)
4. Clinical instability (systolic blood pressure <100 mm Hg or arterial Oxygen saturation <92% at ambient air) at the time of presentation
5. Active bleeding or at high risk of bleeding
6. Severe renal failure (creatinine clearance <30ml/min)
7. Severe liver insufficiency (Child-Pugh B or C)
8. Concomitant use of strong CYP3A4 inhibitors or strong CYP3A4 inducers
9. Known hypersensitivity to rivaroxaban
10. Need for therapeutic anticoagulation for another reason
11. Therapeutic anticoagulation for >72 hours for any reason at the time of screening
12. Hospitalized for >72 hours prior to the diagnosis of isolated SSP (hospital-acquired VTE)
13. Known pregnancy or breast feeding (pregnancy test to be performed for women of childbearing potential)
14. Lack of safe contraception in women of childbearing potential
15. Refusal or inability to provide informed consent
16. Prior enrolment in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Recurrent venous thromboembolism | Within 90 days of randomization
  Proportion of recurrent, clinically symptomatic, objectively confirmed venous thromboembolism (defined as recurrent fatal or nonfatal pulmonary embolism or lower limb deep vein thrombosis)

SECONDARY OUTCOMES:
Clinically significant bleeding | Within 90 days of randomization
  Proportion of the composite of major and clinically relevant non-major bleeding
All-cause mortality | Within 90 days of randomization
  Proportion of deaths (all causes of death will be considered)

OTHER OUTCOMES:
Health-related quality of life | Within 90 days of randomization
  Pulmonary embolism related quality of life as assessed by the Pulmonary Embolism Quality of Life (PEmb-QoL) questionnaire
Functional status | Within 90 days of randomization
  Functional status as assessed by the post-venous thromboembolism functional status scale
Initial length of stay (LOS) | Within 90 days of randomization
  Defined as the time/date of discharge minus time/date of admission at the emergency department
Subsequent overall hospitalizations | Within 90 days of randomization
  Number of overall hospitalizations
Emergency departments and physician outpatient visits | Within 90 days of randomization
  Number of emergency department and physician outpatient visits
Return to work or usual activities | Within 90 days of randomization
  Time (days) to return to work in workers and usual activities (household) in non-workers

CONTACTS AND LOCATIONS:
Overall Officials: Drahomir Aujesky, Prof. MD MSc, Study Director — Inselspital, Bern University Hospital, University of Bern
Locations (39):
- Belgium (2):
  - Centre hospitalier universitaire de Liege, Liège
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
- The Ottawa Hospital, Ottawa, Canada
- France (7):
  - Hôpital Bicêtre - APHP, Le Kremlin-Bicêtre, Le Kremlin-Bicêtre
  - Centre Hospitalier Regional Et Universitaire De Brest, Brest
  - CHU Gabriel-Montpied, Clermont-Ferrand
  - Centre Hospitalier Universitaire De Dijon, Dijon
  - Hospital Edouard Herriot, Lyon
  - CHU De Rouen, Rouen
  - CHU ST Etienne - Hôpital Nord, Saint-Priest-en-Jarez
- Netherlands (6):
  - Albert Schweitzer Ziekenhuis Dordrecht, Dordrecht
  - Medisch Spectrum Twente, Enschede
  - Leiden University Medical Center, Leiden
  - Erasmus Universitair Medisch Centrum, Rotterdam
  - Haaglanden Medisch Centrum, The Hague
  - Isala Klinieken Zwolle, Zwolle
- Switzerland (23):
  - Cantonal Hospital of Liestal, Liestal, Basel
  - Cantonal Hospital of Aarau, Aarau, Canton of Aargau
  - University Hospital Inselspital, Bern, Canton of Bern
  - Hospital of Bienne, Biel/Bienne, Canton of Bern
  - Cantonal Hospital of Fribourg, Fribourg, Canton of Fribourg
  - Cantonal Hospital of Lucerne, Lucerne, Canton of Lucerne
  - Cantonal Hospital of Olten, Olten, Canton of Solothurn
  - Cantonal Hospital of St. Gallen, Sankt Gallen, Canton of St. Gallen
  - University Hospital of Lausanne, Lausanne, Canton of Vaud
  - Hospital of Nyon, Nyon, Canton of Vaud
  - Cantonal Hospital of Winterthur, Winterthur, Canton of Zurich
  - Triemli Hospital, Zurich, Canton of Zurich
  - University Hospital Zürich, Zurich, Canton of Zurich
  - Cantonal Hospital of Frauenfeld, Frauenfeld, Thurgau
  - Hospital of Sion, Sion, Valais
  - Cantonal Hospital of Uri, Altdorf
  - Cantonal Hospital of Baden, Baden
  - University Hospital of Basel, Basel
  - Tiefenau Hospital, Bern
  - Regional Hospital of Emmental, Burgdorf
  - Hospital of Delémont, Delémont
  - Geneva University Hospital, Geneva
  - Hospital of Neuchâtel, Neuchâtel

IPD SHARING:
Plan to Share IPD: Yes
After publication of the study results, a de-identified patient-level data set relating to the primary publication along with the latest version of the study protocol, the informed consent form, the statistical analysis plan, the code used for the analyses, and the Data Management and Quality Plan describing all data management aspects of the study will be made publicly available for replication of the study results and secondary data analyses in the Bern Open Repository and Information System (BORIS) Research Data, an online non-commercial data repository that meets Swiss National Science Foundation requirements for FAIR Data Principles (www.force11.org/group/fairgroup/fairprinciples)
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After publication of the study results
Access Criteria: Data will be publicly available for replication of the study results and secondary data analyses in the Bern Open Repository and Information System (BORIS) Research Data
URL: https://www.boris.unibe.ch/

REFERENCES:
- [Derived] Baumgartner C, Klok FA, Carrier M, Limacher A, Moor J, Righini M, Beer JH, Peluso M, Rakovic D, Huisman MV, Aujesky D. Clinical Surveillance vs. Anticoagulation For low-risk patiEnts with isolated SubSegmental Pulmonary Embolism: protocol for a multicentre randomised placebo-controlled non-inferiority trial (SAFE-SSPE). BMJ Open. 2020 Nov 19;10(11):e040151. doi: 10.1136/bmjopen-2020-040151. PMID 33444199